CLINICAL TRIAL: NCT04698044
Title: Anxiety and Depression Perceived by Individuals With and Without Cancer During the COVID-19 Pandemic Period: A Population-based Comparative Study
Brief Title: Anxiety and Depression Perceived by Individuals With and Without Cancer During the COVID-19 Pandemic Period
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, M.D., Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: COVFAIROFALL
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Depression; Covid19; Cancer; Chronic Disease
Keywords: anxiety; depression; covid-19; cancer; chronic disease
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19; Neoplasms; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Have not chronic disease
  Interventions: Diagnostic Test: Hospital Anxiety Depression Scale
- Cancer: Have cancer
  Interventions: Diagnostic Test: Hospital Anxiety Depression Scale
- Non-Cancer Crhronic Disease: Have non-cancer chronic disease
  Interventions: Diagnostic Test: Hospital Anxiety Depression Scale

INTERVENTIONS:
Diagnostic Test: Hospital Anxiety Depression Scale — HADS is a self-report questionnaire designed to screen the symptoms of anxiety and depression in individuals with medical diseases other than psychiatric illnessesHADS is a self-report questionnaire designed to screen the symptoms of anxiety and depression in individuals with medical diseases other than psychiatric illnesses The 4-point Likert type scale, which consists of 14 items, has 2 subscales. Each of the HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D) subscales has 7 items. The score given for each question varies between 0 and 3. A high score indicates a high level of anxiety and depression. The responses given to the questions are given certain scores, and as a result, a score of 0-7 refers to a normal level, 8-10 to a level at the limit and 11 and above to a high level (abnormal level).

SUMMARY:
The COVID-19 pandemic has negatively affected individuals not only physiologically but also psychologically. The aim of this study is to examine the anxiety and depression status of cancer patients, individuals with non-cancer chronic diseases and healthy individuals with an online screening questionnaire during the COVID-19 pandemic period.

DETAILED DESCRIPTION:
Our aim is to evaluate and compare the anxiety and depression status of cancer patients, individuals with non-chronic chronic diseases and healthy individuals during the COVID-19 period with an online screening program.

A simple random sampling method performed by a computer was used in selecting the participants from 7,000 people whose information was available in the hospital automation system. The computer program enumerates the items in the sampling frame, determines its own random numbers, and presents the selected items to the researcher in writing or digitally (Newman & Ridenour, 1998).

The sample groups were randomly selected from cancer patients, patients with non-cancer chronic diseases and those without any diseases. The study included individuals who were aged 18 years and above, volunteered to participate in the study and were literate. The diagnoses recorded in the electronic medical records of the patients were examined, and those diagnosed with psychiatric diseases (depression, mania, bipolar disorder, psychosis, obsessive-compulsive disorder, etc.), mental retardation, dementia, and Alzheimer's disease were excluded. In addition, the questionnaire questions include the question of the presence of existing psychiatric and neurological diseases. The patient was excluded from the study also if these diagnoses were reported by the patient. Moreover, the participation of the patient in the study was not allowed in the presence of both cancer and a non-cancer chronic disease. Non-cancer chronic diseases were defined as diabetes mellitus, hypertension, neurological diseases, asthma, chronic obstructive pulmonary disease (COPD), other pulmonary diseases, cardiovascular diseases, and hypothyroidism. Other patients who used chronic medication and/or were followed up for any chronic disease (rheumatic disease, endocrinal disorders, liver disease, kidney diseases) were classified as other chronic diseases. Approval was taken from the University of Health Sciences, XXX Ethics Committee (approval number: 20/133) before the study commenced. The patients were called with phone and confirmed whether they wanted to participate in the study, and their consents were obtained. Individuals who wanted to participate in the study was informed about the purpose of the study, procedure and data privacy, and told that participation was on a voluntary basis, and individuals could leave the research at any time they wanted. Individuals read and signed their consent forms online. The study was conducted in compliance with the "Ethical principles for medical research involving human subjects" of the Helsinki Declaration. All data were collected with Survey Monkey (2005 SurveyMonkey.com), which provides electronic self-control, prevents multiple entries from the same person, and makes it easier to collect and track data (last data entry: 07/06/2020). Confidentiality was guaranteed by completely deactivating electronic records and IP address records.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients, patients with non-cancer chronic diseases and those without any diseases
* 18 years or above
* Literate

Exclusion Criteria:

* Psychiatric diseases (depression, mania, bipolar disorder, psychosis, obsessive-compulsive disorder, etc.)
* Mental retardation
* Dementia
* Alzheimer's disease were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample groups were randomly selected from cancer patients, patients with non-cancer chronic diseases and those without any diseases
Sampling Method: Non-Probability Sample
Enrollment: 1107 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
HADS | 14 days
  The score of Hospital Anxiety Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No